CLINICAL TRIAL: NCT04343794
Title: Using Biovitals® Sentinel to Monitor Disease Progression in Subjects Quarantined for Suspected COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ivan FN Hung MD, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COVID19_Biovitals_Protocol_1
Record Dates: First submitted 2020-02-20; First posted 2020-04-13 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: COVID19
Keywords: Wearable physiological monitor
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biovitals (Experimental): Continuous physiological monitoring using Biovitals platform including (1) armband with multiple physiological sensor, (2) remote monitoring, and (3) Analytic platform. The arm will be worn 23 hours a day and off for 1 hour during showering for recharging battery during 24 hr quarantine period
  Interventions: Device: BIOVITALS
- Control (No Intervention): Usual standard care

INTERVENTIONS:
Device: BIOVITALS — Biovitals platform including (1) armband with multiple physiological sensor, (2) remote monitoring, and (3) Analytic platform. The arm will be worn 23 hours a day and off for 1 hour during showering for recharging battery during 24 hr quarantine period
  Arms: Biovitals

SUMMARY:
The novel coronavirus (COVID-19) emerged in December 2019, and in mere months has spread to more than 104 countries, resulting in an outbreak of viral pneumonia worldwide.

Current local quarantine policy in Hong Kong for individuals suspected for COVID-19 requires daily self-reported symptomatology and body temperature, given the intermittent nature and the high dependency of self-discipline undermine the practicality of the approach. To date, the advance in sensor technology has made possible to continuously monitor individual physiological parameters using a simple wearable device. Together with the mobile wearable technology that allowing instantaneous, multi-directional, and massive data transfer, remote continuous physiological monitoring is made possible. The Cardiology division, the Univeristy of Hong Kong has been in collaboration with Biofourmis to implement such technology for remote heart failure management. Similar digital therapeutic system can be applied to remotely monitor physiological parameters of large number of quarantined or suspected COVID-19 at home or in quarantine facility. It is purposed to allow the monitoring team to effectively and remotely monitor COVID-19 quarantined and patients, manage and evaluate the disease progression.

DETAILED DESCRIPTION:
Owing to the massive outbreak of COVID-19, as of March 9, 2020, the virus has reportedly caused 108,618 infections and 3,800 deaths globally. The World Health Organization (WHO) has declared COVID-19 disease a public health emergency of international concern. As there has yet been specific therapeutic or vaccine for the condition, rigorous implementation of traditional public health measures including isolation, quarantine, social distancing, and community containment is the principle strategy to control the COVID-19 epidemic. In addition to the isolation of confirmed COVID-19 infected patients from noninfected population, it is equally if not more important to quarantine asymptomatic individuals with possible exposure to COVID-19 in order to reduce the viral spread. Indeed, quarantine measures have been initiated in many countries and regions, which restrict movements of asymptomatic individuals with COVID-19 exposure often with fever and symptom surveillance at home or designated facilities for the presumed incubation period (14 days). While conceptually attractive, the intermittency and high dependency of selfdiscipline for body temperature and symptom surveillance undermine the practicality and effectiveness of the approach. Furthermore, it has been reported that as many as 50% of COVID-19 infected patients had not had fever until the full-blown disease, thereby body temperature surveillance per se may not be sufficient to detect early disease progression.

In the past few decades, advances in sensor technology miniaturize electronic physiological sensors that could be incorporated into wearable devices allowing continuous monitoring of physiological parameters such as skin temperature, heart rate, respiratory rate, oxygen saturation, perspiration and activity of ambulatory subjects in a 24/7 basis. Together with current telecommunication platform capable of instantaneous and multi-directional massive data transfer, it is possible to remotely monitor a large number of individual subjects' physiological parameters in a real-time manner, and relay to managing physicians for timely intervention. Nonetheless, such potentials have not been fully explored in the real-world disease management. The current study will assess the impact of remote continuous real-time physiological monitoring using wearable armband device Everion® (Biofourmis, Singapore) and artificial intelligence-powered analytical platform Biovitals® Sentinel (Biofourmis, Singapore) on detection of disease progression in asymptomatic subjects with COVID-19 exposure under mandatory quarantine at designated facilities in Hong Kong. The research hypothesis is that by processing continuous physiological data collected using wearable device Everion® and patient reported outcomes with a cloud-based analytics platform Biovitals® Sentinel, it will possible to detect physiological changes and other clinically meaningful alerts that indicate early clinical progression in quarantined subjects with COVID-19 exposure.

The wearable vital sign monitor Everion® is capable to track multiple vitals sings including heart rate, heart rate variability, blood pulse variation, respiration rate under rest, activity, steps, skin temperature and etc. It is Bluetooth connected to a dedicated study-smartphone that allows remote transfer of all the physiological data captured by the wearable device in real time. A specially-designed application (APP) on the study-smartphone enables the patient to participate in health monitoring by reporting symptoms regularly and make aware of his/her physical and physiological patterns via the monitoring displays on the smart-phone. The patient's passive physiological data from the device and the active data on the symptoms and outcomes from Biovitals® analytics platform are automatically transferred to the monitoring console on the cloud. Thus, the Biofourmis platform solution is proposed to allow the monitoring team to effectively and remotely monitor COVID-19 patients and evaluate the disease progression. Leveraging Everion, the smartphone APP, Biovitals® analytics platform and the caregiver dashboard, biofourmis has built an end to end solution, Biovitals® Sentinel to remote monitor and manage the suspected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥18 years of age
* Quarantined as suspected COVID-19
* Asymptomatic upon enrolment
* All subjects give written informed consent

Exclusion Criteria:

- Failure to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Time to diagnosis of COVID-19 by RT-PCR in subjects | within 14 days
  Time from quarantine to diagnosis of COVID-19

SECONDARY OUTCOMES:
Compliance to complete the study | within 14 days
  Adherence to device
Sensitivity and specificity of Biovitals® Sentinel | within 14 days
  To identify COVID19 subjects
Cross infection rate within the family cluster | within 14 days
  % of family members infection
Length of hospital stay of positive subjects | 1 year at study completion
  Length of hospital stay
Length of ICU stay of positive patients | 1 year at study completion
  Length of ICU stay
National Early Warning Score 2 rating of positive patients | 4 weeks from diagnosis
  Vital signs of positive patients
Viral load of positive patients | 4 weeks from diagnosis
  Virology laboratory result of nasopharyngeal swab
Worsening of comorbidities | 1 year at study completion
  Worsening of comorbidities
Mortality | 1 year at study completion
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: David Siu, MD FRCP, Principal Investigator — HKU
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided